CLINICAL TRIAL: NCT02284022
Title: Protocole de Validation Clinique du Logiciel d'Interface Cerveau-Ordinateur RoBIK Pour la Communication Des Patients Atteints de Maladie Neuromusculaires (MNM)
Brief Title: Clinical Validation Protocol for BCI for the Communication of Patients Suffering From Neuromuscular Disorders.
Acronym: PVCAFM
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 14055
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Communication; Neuromuscular Disease
MeSH Terms: conditions — Communication; Neuromuscular Diseases | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brain Computer Interface: Patients will test the brain computer interface system
  Interventions: Device: Brain computer interface

INTERVENTIONS:
Device: Brain computer interface — Recording the P300 Testing the device Using the device with a speller

SUMMARY:
the objective of this protocol is evaluate the safety and tolerance of a communication system for severely disable patients with myopathies. The system analyses the brain electric activity in real time and converts it into digital commands for a spelling device, which is refered to as the P300 speller in the scientific literature. The secondary objective is to compare the performance of such tool with a more traditional assistive technology for the communication of severely disabled patients : scanner systems.

DETAILED DESCRIPTION:
This is a pilot study for which 15 patients with myopathies will be included. The primary objective of the study is to assess the safety and tolerance of a system for communication named P300 speller. The P3Speller is a brain computer interface (BCI) that records the brain electric activity with the use of electroencephalography (EEG) and analyzes it in real time in order to identify slight changes generated in relation to a visual stimulation (evoked potentials). The identification of such brain potentials is translated into a digital command for a spelling device. The secondary objective of this study is to compare the efficacy of this spelling device with a more traditional assisitve technology called scanner interface. A scanner interface uses single clicks that can be obtaines with an adequate interface which exploits the remaining muscular activity from a patients.

Every patient will use each interface (P300 sepller and Scanning) with a randomized order. Results will bec o,pared in terms of information flow from the patient to the computer expressed in bit rate per minute.

ELIGIBILITY:
Inclusion Criteria:

* Adult older than 18y.o., diagnosed with neuromuscular disease, stable vital signs and informed consent

Exclusion Criteria:

* History of seizure, brain damage, sight or auditory dysfunction, Atopic dermatitis, skin hypersensitivity to gold, patient under guardianship, illiterates or not able to cooperate , cognitive dysfunction
* Steinert disease, Merosine negative disease, Alpha-dystroglycanopathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: neuromuscular disease patients
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Bit rate (BR) the amount fo information that flows from the patient to the computer during the spelling session. This criterion is a combination of the number of symbols selected, the accuracy, and the time. | 30 minutes
  The comparison criteria for performance was the bitrate, br, that is defined by (Wolpow et al. 2000):
  〖br=log〗_2 (M)+p.log_2 p+(1-p) 〖log〗_2 (1-p)/(M-1) where M=36 is the number of symbols p the spelling accuracy (the percentage of correctly identified symbols).

SECONDARY OUTCOMES:
patient satisfaction (visual analogic scale) | 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: David Orlikowski, MDPhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital R. Poincaré, Garches, France

IPD SHARING:
Plan to Share IPD: Undecided